CLINICAL TRIAL: NCT02890771
Title: To Evaluate the Efficacy of Whole Turmeric Powder in Gingival Massaging and as an Adjunct to Scaling and Root Planing in Patients With Chronic Periodontitis
Brief Title: Efficacy of Turmeric in Gingival Massaging and Adjunct to Scaling and Root Planing in Chronic Periodontitis Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Government College of Dentistry, Indore (Other)
Responsible Party: Principal Investigator, SAURABH KUMAR DUBEY, Post graduate student, Government College of Dentistry, Indore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GDCHIndore
Record Dates: First submitted 2016-09-01; First posted 2016-09-07 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Chronic Periodontitis
Keywords: Turmeric; Chronic periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Toothbrushing; Dentifrices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tooth Brushing (Active Comparator): Tooth brushing with dentifrice
  Interventions: Procedure: Turmeric Massaging; Procedure: SRP with turmeric massaging
- Turmeric massaging (Experimental): Tooth Brushing,massaging with whole turmeric powder
  Interventions: Procedure: Tooth Brushing with Dentifrice; Procedure: SRP with turmeric massaging
- SRP with turmeric massaging (Experimental): SRP with turmeric massaging on half arch
  Interventions: Procedure: Tooth Brushing with Dentifrice; Procedure: Turmeric Massaging

INTERVENTIONS:
Procedure: Tooth Brushing with Dentifrice — Tooth Brushing with Dentifrice (Standard Tooth Brushing technique will be demonstrated by using same type of tooth brush and toothpaste).
  Arms: SRP with turmeric massaging; Turmeric massaging
Procedure: Turmeric Massaging — :-Tooth Brushing with Dentifrice (with same type of tooth brush and toothpaste) and massaging with whole Turmeric Powder.
  Arms: SRP with turmeric massaging; Tooth Brushing
Procedure: SRP with turmeric massaging — on one side of the arch only Scaling and Root Planing(SRP) to be done, while on the other side, after the Scaling and Root Planing massaging with whole Turmeric Powder shall be carried out by the patients/subjects
  Arms: Tooth Brushing; Turmeric massaging

SUMMARY:
Periodontal disease is considered as inflammatory, multifactorial, and threshold disease accompanied by destruction of periodontium and eventually the loss of natural teeth. Periodontal disease is highly prevalent dental disease especially, in developing and underdeveloped countries affecting more or less 80% of the population. For the prevention of this highly prevalent dental affliction, still no effective and practical preventive measures are available which can reduce its high prevalence rate though, lot of research work is going on.

DETAILED DESCRIPTION:
Various interceptive and therapeutic modalities are available comprising of non-surgical and surgical therapies. But, these therapies are not available for everyone, due to various reasons such as low socio-economic conditions of the majority of the population including poverty, illiteracy, and malnutrition etc. along with low dentist: population ratio. Moreover, the availability of a dentist and/or periodontist is limited in rural and remote areas, whereas the prevalence rate of periodontal disease is comparatively higher in these areas than that of urban areas.

Looking to these difficulties, the investigators have to think and explore the beneficial effects by conducting research work on various home care measures which are being used since many generations, especially in our country and thus people were/are enjoying the benefits with almost all or many natural teeth, up to last span of their lives.Though, the scientific evidences of beneficial effects of home care measures for cleaning and massaging of teeth and gums, respectively are not yet evident significantly. But, traditional uses of various dentifrices those are still in practices and thus need scientific attentions. Now, the investigators are in the evidence based era, especially in the field of medical sciences. Therefore, the number of research studies should be planned and carried out at various centres in different parts of the country, to ascertain the beneficial effects of traditional oral hygiene practices such as: Datoons (Neem, Babool etc), leaves of various plants like Mango, Charcoal powder, Meswak, salt, Mustard oil with Salt, and Turmeric powder and other such home care dental cleansing materials. After getting the beneficial information's/evidences accordingly, the uses of specific traditional materials and methods for the cleansing of the teeth and massaging of the gums can be advocated. And thus, specifically the developing and underdeveloped countries may be benefitted.

Out of various home care dental cleansing materials the Turmeric powder is not only being used as one of important condiments of our kitchen, and at the same time as a medicinal use since ages.

The 'Turmeric' is known for its anti-inflammatory, antioxidant, antimicrobial, immune stimulant, antiseptic, anti-carcinogenic, and anti-mutagenic properties [1]. Drake [2] and Han et al [3], observed anti- microbial activity of Turmeric. Roobal Bahal et al [4] stated that on use of 2% Turmeric gel, significant reduction in the mean plaque index, gingival index, sulcus bleeding index, probing pocket depth and significant reduction in trypsin like enzymatic activity of "Red-Complex" microorganisms. Ruchika Jaswal et al [5] conducted a pilot study to evaluate and compare the clinical effects of topical subgingival application of 2% whole turmeric gel and 1% chlorhexidine gel as an adjunct to scaling and root planing (SRP) in patients suffering from chronic periodontitis.

Very few studies, which can be counted on fingers, have been conducted worldwide in this direction. Hence, this study is being taken to evaluate the efficacy of whole Turmeric Powder in Gingival Massaging and as an adjunct to Scaling and Root Planing in Patients with Chronic Periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* Cases with moderate to severe form of Generalized Chronic Periodontitis patients of any sex.
* Patients in the age group of 35-65 years, who abide by approved protocol guidelines, and are ready to give written informed consent.

Exclusion Criteria:

* Any known systemic disease which has effects on periodontium such as diabetes etc.
* Patients on anti-inflammatory, antibiotics and perioceutics, since 3 months.
* Patients who have known allergy to material used for the study.
* Pregnant and lactating mothers.
* Patients had undergone any kind of non-surgical and/or surgical periodontal therapy earlier, in past 6 months.
* Tobacco users.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Plaque Index (Turesky modification of Quigley Hein Index, 1970) | baseline

SECONDARY OUTCOMES:
Plaque Index (Turesky modification of Quigley Hein Index, 1970) | 1 week
Plaque Index (Turesky modification of Quigley Hein Index, 1970) | 2 week
Plaque Index (Turesky modification of Quigley Hein Index, 1970) | 4 week
Plaque Index (Turesky modification of Quigley Hein Index, 1970) | 6 week
Gingival Index (Loe H and Silness J 1963) | baseline
Gingival Index (Loe H and Silness J 1963) | 1 week
Gingival Index (Loe H and Silness J 1963) | 2 week
Gingival Index (Loe H and Silness J 1963) | 4 week
Gingival Index (Loe H and Silness J 1963) | 6 week
Russell's Periodontal Index (Rusell's A.L, 1956) | baseline
Russell's Periodontal Index (Rusell's A.L, 1956) | 1 week
Russell's Periodontal Index (Rusell's A.L, 1956) | 2 week
Russell's Periodontal Index (Rusell's A.L, 1956) | 4 week
Russell's Periodontal Index (Rusell's A.L, 1956) | 6 week
Periodontal Probing Depth | baseline
Periodontal Probing Depth | 1 week
Periodontal Probing Depth | 2 week
Periodontal Probing Depth | 4 week
Periodontal Probing Depth | 6 week
Clinical Attachment Levels | baseline
Clinical Attachment Levels | 1 week
Clinical Attachment Levels | 2 week
Clinical Attachment Levels | 4 week
Clinical Attachment Levels | 6 week

CONTACTS AND LOCATIONS:
Overall Officials: Dr Subhash Garg, MDS, Study Chair — Govt. Dental College, Indore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Izui S, Sekine S, Maeda K, Kuboniwa M, Takada A, Amano A, Nagata H. Antibacterial Activity of Curcumin Against Periodontopathic Bacteria. J Periodontol. 2016 Jan;87(1):83-90. doi: 10.1902/jop.2015.150260. Epub 2015 Oct 8. PMID 26447754
- [Background] Farjana HN, Chandrasekaran SC, Gita B. Effect of oral curcuma gel in gingivitis management - a pilot study. J Clin Diagn Res. 2014 Dec;8(12):ZC08-10. doi: 10.7860/JCDR/2014/8784.5235. Epub 2014 Dec 5. PMID 25654020
- [Background] Zhou T, Chen D, Li Q, Sun X, Song Y, Wang C. Curcumin inhibits inflammatory response and bone loss during experimental periodontitis in rats. Acta Odontol Scand. 2013 Mar;71(2):349-56. doi: 10.3109/00016357.2012.682092. Epub 2012 May 4. PMID 22554269